CLINICAL TRIAL: NCT00482040
Title: Randomized Trial Investigating Four Nasal CPAP Systems in the Management of Apnea of Prematurity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting took longer than expected due to a lack of eligible patients (very strong inclusion and exclusion criterias)
Sponsor: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CPAP-I-Study
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2007-08-24 (Estimated); Status verified 2007-05

CONDITIONS: Continuous Positive Airway Pressure; Apnea of Prematurity; CPAP
Keywords: CPAP; Preterm; Prematurity; Apnea of prematurity
MeSH Terms: conditions — Apnea; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Stephanie (TM), Infant Flow (TM), Infant Flow advance (TM), Bubble CPAP

SUMMARY:
The purpose of this study is to evaluate four different nasal continuous pressure systems, which are usually applied on our neonatal intensive care unit, with regard of their effect on bradycardia and desaturations in preterm infants.

DETAILED DESCRIPTION:
BACKGROUND:

Apnea of prematurity (AOP) is a common problem in preterm infants. Nasal respiratory support using either Continuous Positive Airway Pressure (CPAP) or Intermittent Mandatory Ventilation (IMV) are, among others, widely used treatments. Which of the different systems is the most efficient, however, is unclear.

OBJECTIVE:

Efficiency of different CPAP systems on reducing the cumulative percentage of bradycardia and desaturation in preterm infants.

METHODS:

In a prospective, randomized, cross-over trial 32 preterm infants Infants will randomly allocated to receive nasal CPAP delivered by one of the following sys-tems: (1) a conventional IMV-System (Stephanie, Stephan GmbH, Germany with PIP 15 cmH2O, RR 10/min) delivering CPAP via short binasal prongs (Hudson RCI, USA); (2) the Infant-Flow-System (EME Ltd, Great Britain) with CPAP delivery via short binasal prongs; (3) the Infant-Flow-AdvanceTM-System used in the pressure assist mode with PIP 10 cmH2O, RR 10/min; and (4) a nasal underwater bubble CPAP with application via binasal prongs (Hudson RCI, USA).

All systems will be adjusted to achieve an approximate PEEP of 6 cm H2O. Each study lasts 24 hours, during which chest wall and abdominal movements, SaO2, tcPCO2, ECG, esopha-gus pressure and CPAP-/IMV-pressure will be recorded continuously. Infants will be studied in room air in a 15° head tilt prone position while being treated with caffeine (3mg/kg/d).

PRIMARY OUTCOME MEASURE Cumulative percentage of bradycardia (heart rate <80/min) and desaturation (SaO2 <80%) per hour.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at birth < 34 weeks
* postconceptional age and body weight at study ≤38 week and >1000 g
* requirement for N-CPAP to treat AOP as judged by the attending neonatologist

Exclusion Criteria:

* congenital or chromosomal abnormalities
* acute infections
* intraventricular hemorrhage
* additional inspired oxygen to maintain pulse oximeter saturation SpO2 >92%
* patent ductus arteriosus

Max Age: 14 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2004-03; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Cumulative percentage of bradycardia (heart rate <80 beats/min) and desaturation (SaO2 <80%) per hour | one year

SECONDARY OUTCOMES:
- Event rates for central apneas, desaturations and bradycardias calculated as the number of respective events per hour of artefact free recording time - relative cumulative event time - baseline heart rate, respiratory rate and oxygen saturation | one year

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Pantalitschka, MD, Principal Investigator — University children´s hospital Tuebingen